CLINICAL TRIAL: NCT00985959
Title: A Phase I/II Clinical Study of JNJ-26866138 (Bortezomib) in Untreated Multiple Myeloma Patients Who Are Not Candidates for Hematopoietic Stem Cell Transplant (HSCT)
Brief Title: A Study of JNJ-26866138 (Bortezomib) in Untreated Multiple Myeloma Patients Who Are Not Candidates for Hematopoietic Stem Cell Transplant (HSCT)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR014776; JNJ-26866138-JPN-MM-102 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2009-09-18; First posted 2009-09-29 (Estimated); Results first posted 2013-12-02 (Estimated); Last update posted 2013-12-02 (Estimated); Status verified 2013-10

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; Hematopoietic stem cell transplant; HSCT; Melphalan; Prednisolone; Bortezomib; JNJ-26866138
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Melphalan; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Phase I: JNJ-26866138 0.7 mg/m2 (Experimental): JNJ-26866138 0.7 mg/m2 on Days 1, 4, 8, 11, 22, 25, 29 and 32 of 6-week cycle up to 4 cycles. Melphalan 9 mg/m2 and Prednisolone 60 mg/m2 on Days 1, 2, 3 and 4 of 6-week cycle up to 4 cycles.
  Interventions: Drug: JNJ-26866138 0.7 mg/m2; Drug: Melphalan; Drug: Prednisolone
- Phase I: JNJ-26866138 1.0 mg/m2 (Experimental): JNJ-26866138 1.0 mg/m2 on Days 1, 4, 8, 11, 22, 25, 29 and 32 of 6-week cycle up to 4 cycles. Melphalan 9 mg/m2 and Prednisolone 60 mg/m2 on Days 1, 2, 3 and 4 of 6-week cycle up to 4 cycles
  Interventions: Drug: JNJ-26866138 1.0 mg/m2; Drug: Melphalan; Drug: Prednisolone
- Phase I: JNJ-26866138 1.3 mg/m2 (Experimental): JNJ-26866138 1.3 mg/m2 on Days 1, 4, 8, 11, 22, 25, 29 and 32 of 6-week cycle up to 4 cycles. Melphalan 9 mg/m2 and Prednisolone 60 mg/m2 on Days 1, 2, 3 and 4 of 6-week cycle up to 4 cycles
  Interventions: Drug: JNJ-26866138 1.3 mg/m2; Drug: Melphalan; Drug: Prednisolone
- Phase II: JNJ-26866138 1.3 mg/m2 (Experimental): JNJ-26866138 1.3 mg/m2 on Days 1, 8, 22 and 29 of 6-week cycle for 5-9 cycles. Melphalan 9 mg/m2 and Prednisolone 60 mg/m2 on Days 1, 2, 3 and 4 of 6-week cycle up to 9 cycles
  Interventions: Drug: JNJ-26866138 1.3 mg/m2; Drug: Melphalan; Drug: Prednisolone

INTERVENTIONS:
Drug: JNJ-26866138 0.7 mg/m2 — JNJ-26866138 0.7 mg/m2 will be administered intravenously on Days 1, 4, 8, 11, 22, 25, 29 and 32 of 6-week cycle up to 4 cycles.
  Other Names: bortezomib
  Arms: Phase I: JNJ-26866138 0.7 mg/m2
Drug: JNJ-26866138 1.0 mg/m2 — JNJ-26866138 1.0 mg/m2 will be administered intravenously on Days 1, 4, 8, 11, 22, 25, 29 and 32 of 6-week cycle up to 4 cycles
  Other Names: bortezomib
  Arms: Phase I: JNJ-26866138 1.0 mg/m2
Drug: JNJ-26866138 1.3 mg/m2 — Phase I: JNJ-26866138 1.3 mg/m2 will be administered intravenously on Days 1, 4, 8, 11, 22, 25, 29 and 32 of 6-week cycle up to 4 cycles. Phase II: JNJ-26866138 1.3 mg/m2 on Days 1, 8, 22 and 29 of 6-week cycle for 5 to 9 cycles.
  Other Names: bortezomib
  Arms: Phase I: JNJ-26866138 1.3 mg/m2; Phase II: JNJ-26866138 1.3 mg/m2
Drug: Melphalan — Melphalan 9 mg/m2 will be taken orally (by mouth) on Days 1, 2, 3 and 4 of 6-week cycle up to 9 cycles
Drug: Prednisolone — Prednisolone 60 mg/m2 will be taken orally (by mouth) on Days 1, 2, 3 and 4 of 6-week cycle up to 9 cycles

SUMMARY:
The purpose of the study in Phase I is to select the recommended dose of bortezomib in combination with melphalan and prednisolone in Japanese participants. In Phase II, to assess the effectiveness and safety of the recommended dose of bortezomib (selected in the phase I portion).

DETAILED DESCRIPTION:
This is an open-label (both physician and participant know the intervention), non-randomized (participants are not assigned by chance), multi-center study in untreated multiple myeloma participants who were not candidates for hematopoietic stem cell transplant. This study consists of two parts: Phase I and Phase II. In Phase I, a total of 18 participants will be enrolled ie, 6 patients per dose level (0.7, 1.0 and 1.3 mg/m2) to determine the recommended dose of bortezomib. In Phase II, additional 83 participants will be enrolled. Safety evaluations will include assessment of adverse events, clinical laboratory test, specifically hematological toxicities.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with symptomatic or nonsecretory multiple myeloma
* Participants who have not received chemotherapy and are not hematopoietic stem cell transplantation candidates
* Participants with a measurable lesion
* Life expectancy greater than or equal to 3 months

Exclusion Criteria:

* Previously received treatment for Multiple Myeloma
* Greater than or equal to Grade 2 peripheral neuropathy or neuropathic pain
* Myocardial infarction within 6 months prior to enrollment or uncontrolled angina, severe uncontrolled ventricular arrhythmias, or clinically significant conduction system abnormalities
* Patient is known to be seropositive for the human immunodeficiency virus (HIV), Hepatitis B surface antigen-positive or active hepatitis C infection
* Active prior malignancy diagnosed within the last 5 years
* Female participant who is pregnant or breast-feeding
* Participant is enrolled in another clinical research study and/or is receiving an investigational agent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2008-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (28):
- Japan (28):
  - Fukuoka
  - Hiroshima
  - Hitachi
  - Isehara
  - Kamogawa
  - Kanazawa
  - Kawagoe
  - Kobe
  - Kōtoku
  - Kumamoto
  - Kurashiki
  - Kurume
  - Kyoto
  - Nagasaki
  - Nagoya
  - Narita
  - Niigata
  - Okayama
  - Ōsaka-sayama
  - Sapporo
  - Shibukawa
  - Suita
  - Tokushima
  - Tokyo
  - Toyama
  - Toyohashi
  - Utsunomiya
  - Yokohama

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total 101 participants (Phase I: 18 and Phase II: 83) were enrolled at multiple sites in Japan.
Pre-assignment Details: 18 participants were enrolled and treated in Phase I. Total 89 participants were enrolled in Phase II (including 6 participants receiving 1.3 mg/m2 in the Phase I part). Of the 89 participants, 87 were received at least 1 dose of study medication. 2 participants were not treated.
Groups:
- Phase I - JNJ-26866138 0.7 mg/m2 Group: JNJ-26866138 0.7 mg/m2 on Days 1, 4, 8, 11, 22, 25, 29 and 32 of 6-week cycle up to 4 cycles. Melphalan 9 mg/m2 and Prednisolone 60 mg/m2 on Days 1, 2, 3 and 4 of 6-week cycle up to 4 cycles
- Phase I - JNJ-26866138 1.0 mg/m2 Group: JNJ-26866138 1.0 mg/m2 on Days 1, 4, 8, 11, 22, 25, 29 and 32 of 6-week cycle up to 4 cycles. Melphalan 9 mg/m2 and Prednisolone 60 mg/m2 on Days 1, 2, 3 and 4 of 6-week cycle up to 4 cycles
- Phase I and II - JNJ-26866138 1.3 mg/m2 Group: Phase I: JNJ-26866138 1.3 mg/m2 on Days 1, 4, 8, 11, 22, 25, 29 and 32 of 6-week cycle up to 4 cycles. Melphalan 9 mg/m2 and Prednisolone 60 mg/m2 on Days 1, 2, 3 and 4 of 6-week cycle up to 4 cycles. Phase II: JNJ-26866138 1.3 mg/m2 on Days 1, 8, 22 and 29 of 6-week cycle for 5-9 cycles. Melphalan 9 mg/m2 and Prednisolone 60 mg/m2 on Days 1, 2, 3 and 4 of 6-week cycle up to 9 cycles
Period: Overall Study
Arm/Group | Phase I - JNJ-26866138 0.7 mg/m2 Group | Phase I - JNJ-26866138 1.0 mg/m2 Group | Phase I and II - JNJ-26866138 1.3 mg/m2 Group
Started | 6 (Number of participants treated) | 6 (Number of participants treated) | 87 (Number of participants treated)
Completed | 3 (Completed all 9 cycles) | 3 (Completed all 9 cycles) | 28
Not Completed | 3 | 3 | 59
Not completed — Adverse Event | 0 | 0 | 19
Not completed — Withdrawal by Subject | 0 | 0 | 8
Not completed — Progressive disease | 1 | 2 | 8
Not completed — Unrecovered toxicity | 0 | 0 | 7
Not completed — Pneumonitis or pulmonary fibrosis | 2 | 0 | 2
Not completed — Complete response observed over 2 cycles | 0 | 1 | 4
Not completed — Other | 0 | 0 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I - JNJ-26866138 0.7 mg/m2 Group | Phase I - JNJ-26866138 1.0 mg/m2 Group | Phase I and II - JNJ-26866138 1.3 mg/m2 Group | Total
Number analyzed (Participants) | 6 | 6 | 87 | 99
Age Continuous [Mean (Standard Deviation); unit: Years] | 72.7 (9.2) | 68.5 (6.47) | 70.9 (5.68) | 70.9 (5.94)
Age, Customized [Number; unit: Participants]
  <65 years | 1 | 1 | 3 | 5
  >= 65 and <= 74 years | 2 | 5 | 60 | 67
  >=75 years | 3 | 0 | 24 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 51 | 57
  Male | 3 | 3 | 36 | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicity During the Phase I (Cycle 1)
Description: Dose limiting toxicity defined as an adverse event or adverse drug reaction experienced by the participants during 6 weeks of treatment Cycle 1
Time Frame: 6 weeks
Population: Dose Limiting Toxicity set, Which includes all 18 participants in the Phase I
Measure: Number; unit: Participants
Groups:
- Phase I - JNJ-26866138 1.3 mg/m2 Group: JNJ-26866138 1.3 mg/m2 on Days 1, 4, 8, 11, 22, 25, 29 and 32 of 6-week cycle up to 4 cycles. Melphalan 9 mg/m2 and Prednisolone 60 mg/m2 on Days 1, 2, 3 and 4 of 6-week cycle up to 4 cycles
Arm/Group | Phase I - JNJ-26866138 0.7 mg/m2 Group | Phase I - JNJ-26866138 1.0 mg/m2 Group | Phase I - JNJ-26866138 1.3 mg/m2 Group
Number analyzed (Participants) | 6 | 6 | 6
Participants | 0 | 0 | 1

2. Primary Outcome: Number of Participants With Overall Response (Complete Response [CR] + Partial Response [PR]) - Phase I and II
Description: Response is evaluated as per the criteria for evaluating disease response and progression in patients with multiple myeloma treated by high-dose therapy and haemopoietic stem cell transplantation (Blade et al. 1998). CR: disappearance of the original monoclonal protein from the blood and urine and <5% plasma cells in the bone marrow on at least 2 determinations for a minimum of 6 weeks; no increase in the size or number of lytic bone lesions; disappearance of soft tissue plasmacytomas for at least 6 weeks. PR: ≥50% reduction in the level of serum monoclonal protein for at least 2 determinations 6 weeks apart; If present, reduction in 24-hour urinary light chain excretion by either ≥90% or to <200 mg for at least 2 determinations 6 weeks apart; ≥50% reduction in the size of soft tissue plasmacytomas for at least 6 weeks; no increase in size or number of lytic bone lesions
Time Frame: 54 weeks
Population: Full analysis set: All participants who received at least one dose of the study medication.
Measure: Number; unit: Participants
Groups:
- Phase II - JNJ-26866138 1.3 mg/m2 Group: JNJ-26866138 1.3 mg/m2 on Days 1, 8, 22 and 29 of 6-week cycle for 5-9 cycles. Melphalan 9 mg/m2 and Prednisolone 60 mg/m2 on Days 1, 2, 3 and 4 of 6-week cycle up to 9 cycles
- Total: Participants from both Phase I and Phase II
Arm/Group | Phase I - JNJ-26866138 0.7 mg/m2 Group | Phase I - JNJ-26866138 1.0 mg/m2 Group | Phase I - JNJ-26866138 1.3 mg/m2 Group | Phase II - JNJ-26866138 1.3 mg/m2 Group | Total
Number analyzed (Participants) | 6 | 6 | 5 | 86 | 98
Participants | 6 [54.1 to 100.0] | 5 [35.9 to 99.6] | 4 [28.4 to 99.5] | 60 [58.9 to 79.2] | 71
Statistical Analysis 1: Comparison: Phase II - JNJ-26866138 1.3 mg/m2 Group; Test type: Superiority or Other; p < 0.0001, Binominal test — Significance level 5% one-tailed. Threshold response rate 35%; Overall response rate (%) = 69.8, 95% CI 2-sided [58.9 to 79.2], Standard Error of Mean 4.9

3. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Bortezomib (JNJ-26866138 Alone) - Phase I
Description: Cmax of bortezomib following intravenous administration of JNJ-26866138 at dose of 0.7, 1.0, and 1.3 mg/m2 on Cycle 1/Day 25 (JNJ-26866138 alone)
Time Frame: Day 25 of Cycle 1
Population: Pharmacokinetics-evaluable population: 16 participants were included in pharmacokinetics-evaluable population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase I - JNJ-26866138 0.7 mg/m2 Group | Phase I - JNJ-26866138 1.0 mg/m2 Group | Phase I - JNJ-26866138 1.3 mg/m2 Group
Number analyzed (Participants) | 6 | 6 | 4
ng/mL | 45.43 (10.087) | 59.42 (18.89) | 120.3 (24.527)

4. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Bortezomib (JNJ-26866138 in Combination With Melphalan and Prednisolone) - Phase I
Description: Cmax of bortezomib following intravenous administration of JNJ-26866138 at dose of 0.7, 1.0, and 1.3 mg/m2 on Cycle 2/Day 4 (combination with melphalan and prednisolone)
Time Frame: Day 4 of Cycle 2
Population: Pharmacokinetics-evaluable population: 14 participants were included in pharmacokinetics-evaluable population during Cycle 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase I - JNJ-26866138 0.7 mg/m2 Group | Phase I - JNJ-26866138 1.0 mg/m2 Group | Phase I - JNJ-26866138 1.3 mg/m2 Group
Number analyzed (Participants) | 6 | 5 | 3
ng/mL | 34.40 (5.7986) | 69.50 (19.455) | 88.87 (19.568)

5. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Melphalan - Phase I
Description: Cmax of melphalan at dose of 9 mg/m2 on Cycle 2/Day 4
Time Frame: Day 4 of Cycle 2
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Melphalan: Melphalan 9 mg/m2 on day 1, 2, 3 and 4 of 6-week cycle up to 9 cycles
Arm/Group | Melphalan
Number analyzed (Participants) | 14
ng/mL | 100.2 (49.515)

6. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Prednisolone - Phase I
Description: Cmax of Prednisolone at dose of 60 mg/m2 on Cycle 2/Day 4
Time Frame: Day 4 of Cycle 2
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Prednisolone: Prednisolone 60 mg/m2 on day 1, 2, 3 and 4 of 6-week cycle up to 9 cycles
Arm/Group | Prednisolone
Number analyzed (Participants) | 14
ng/mL | 1131 (223.92)

7. Secondary Outcome: Median Time to First Response - Phase II
Description: Time to first response is the duartion of time required to achieve first response to treatment
Time Frame: up to 54 weeks
Population: Full analysis set: All participants who received at least one dose of the study medication.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Phase II - JNJ-26866138 1.3 mg/m2 Group
Number analyzed (Participants) | 86
Days | 51 [43 to 82]

ADVERSE EVENTS:
Time Frame: 54 weeks
Description: 87 participants who received at least 1 dose of study medication were evaluated for safety.
Arm/Group | Phase I - JNJ-26866138 0.7 mg/m2 Group | Phase I - JNJ-26866138 1.0 mg/m2 Group | Phase I - JNJ-26866138 1.3 mg/m2 Group | Phase II - JNJ-26866138 1.3 mg/m2 Group
Serious Adverse Events (participants affected / at risk) | 2/6 | 2/6 | 1/6 | 29/87
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 6/6 | 87/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I - JNJ-26866138 0.7 mg/m2 Group (N=6) | Phase I - JNJ-26866138 1.0 mg/m2 Group (N=6) | Phase I - JNJ-26866138 1.3 mg/m2 Group (N=6) | Phase II - JNJ-26866138 1.3 mg/m2 Group (N=87)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster dissemin (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prinzmetal angina (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I - JNJ-26866138 0.7 mg/m2 Group (N=6) | Phase I - JNJ-26866138 1.0 mg/m2 Group (N=6) | Phase I - JNJ-26866138 1.3 mg/m2 Group (N=6) | Phase II - JNJ-26866138 1.3 mg/m2 Group (N=87)
Nasopharyngitis (Infections and infestations) | 2 | 1 | 0 | 14
Neutropenic infection (Infections and infestations) | 0 | 1 | 1 | 10
Leukopenia (Blood and lymphatic system disorders) | 6 | 6 | 6 | 86
Lymphopenia (Blood and lymphatic system disorders) | 6 | 6 | 6 | 86
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 6 | 5 | 86
Neutropenia (Blood and lymphatic system disorders) | 6 | 6 | 6 | 84
Anaemia (Blood and lymphatic system disorders) | 2 | 4 | 4 | 60
Leukocytosis (Blood and lymphatic system disorders) | 3 | 2 | 4 | 44
Decreased appetite (Metabolism and nutrition disorders) | 5 | 2 | 5 | 50
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 3 | 4 | 45
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 4 | 43
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 42
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 2 | 4 | 40
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 4 | 1 | 31
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 35
Hyperchloraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 21
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 42
Insomnia (Psychiatric disorders) | 1 | 2 | 2 | 23
Neuropathy peripheral (Nervous system disorders) | 3 | 2 | 5 | 45
Dysgeusia (Nervous system disorders) | 2 | 1 | 1 | 16
Dizziness (Nervous system disorders) | 0 | 1 | 3 | 15
Headache (Nervous system disorders) | 1 | 0 | 2 | 8
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 14
Infection (Infections and infestations) | 0 | 0 | 0 | 8
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 7
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 7
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 5
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 5
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 8
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 2 | 1 | 34
Hypercreatininaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 15
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 7
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 6
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 6
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 5
Peripheral motor neuropathy (Psychiatric disorders) | 0 | 1 | 1 | 7
Somnolence (Psychiatric disorders) | 1 | 0 | 0 | 5
Cataract (Eye disorders) | 0 | 1 | 0 | 4
Hypotension (Vascular disorders) | 1 | 1 | 1 | 13
Hot flush (Vascular disorders) | 1 | 0 | 0 | 7
Hypertension (Vascular disorders) | 0 | 0 | 0 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 6
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 5
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 6
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 5
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 6 | 56
Constipation (Gastrointestinal disorders) | 4 | 2 | 5 | 45
Nausea (Gastrointestinal disorders) | 1 | 2 | 6 | 48
Vomiting (Gastrointestinal disorders) | 0 | 1 | 5 | 36
Stomatitis (Gastrointestinal disorders) | 2 | 2 | 2 | 18
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0 | 1 | 8
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 2 | 9
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 6
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 6
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 5
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 5
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 4
Hepatic function abnormal (Hepatobiliary disorders) | 3 | 1 | 3 | 44
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 6
Rash (Skin and subcutaneous tissue disorders) | 2 | 4 | 3 | 56
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 11
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 10
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 8
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 8
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 4
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 12
Azotaemia (Renal and urinary disorders) | 0 | 1 | 0 | 12
Malaise (General disorders) | 2 | 3 | 5 | 37
Pyrexia (General disorders) | 2 | 1 | 6 | 30
Fatigue (General disorders) | 0 | 1 | 1 | 23
Oedema (General disorders) | 1 | 1 | 2 | 19
Oedema peripheral (General disorders) | 0 | 0 | 2 | 11
Pain (General disorders) | 2 | 2 | 2 | 6
Chest pain (General disorders) | 0 | 0 | 1 | 8
Face oedema (General disorders) | 0 | 1 | 0 | 4
Injection site reaction (General disorders) | 0 | 0 | 0 | 5
C-reactive protein increased (Investigations) | 2 | 3 | 4 | 57
Blood lactate dehydrogenase increased (Investigations) | 0 | 4 | 2 | 50
Weight decreased (Investigations) | 2 | 1 | 2 | 49
Blood alkaline phosphatase increased (Investigations) | 4 | 1 | 1 | 40
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1 | 27
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 2 | 22
Weight increased (Investigations) | 1 | 1 | 2 | 20
Blood urea increased (Investigations) | 0 | 1 | 0 | 11
Blood albumin decreased (Investigations) | 0 | 1 | 0 | 4
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 5
Blood urea decreased (Investigations) | 0 | 0 | 0 | 5
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 6
Blood uric acid decreased (Investigations) | 0 | 0 | 0 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days